CLINICAL TRIAL: NCT01873989
Title: Testosterone Replacement for Male Opioid Agonist Maintained Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1105008492
Record Dates: First submitted 2013-05-22; First posted 2013-06-10 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Chronic Pain; Opioid Addiction; Symptomatic Hypogonadism
Keywords: Chronic pain; Opioid addiction; Symptomatic hypogonadism; Testosterone replacement; Opioid agonist maintenance; Methadone; Buprenorphine
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone replacement (Experimental): Testosterone replacement for hypogonadism.
  Interventions: Drug: Testosterone replacement
- Waitlist control (Other): This arm involves watchful waiting.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Drug: Testosterone replacement
  Arms: Testosterone replacement
Other: Waitlist control
  Arms: Waitlist control

SUMMARY:
This study is designed to develop an effective treatment intervention for chronic pain, symptomatic hypogonadism, and opioid addiction

DETAILED DESCRIPTION:
This study aims to assess the initial efficacy of testosterone replacement in male opioid agonist patients with symptomatic hypogonadism and chronic pain.

The study has two specific aims:

1. To estimate, in male opioid agonist maintained patients, the prevalence of (a)symptomatic hypogonadism and (b) co-occurring symptomatic hypogonadism and chronic pain.
2. To conduct a pilot randomized clinical trial to obtain data regarding the feasibility, acceptability, and efficacy (compared to waitlist control) of testosterone replacement for male patients with chronic pain and opioid dependence, and symptomatic hypogonadism treated with opioid agonist maintenance treatment (N=40).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age
* Male buprenorphine- or methadone-maintained patients at the APT Foundation
* Moderate to severe chronic pain
* Meet criteria for symptomatic hypogonadism
* Understand English
* Interested in receiving testosterone replacement

Exclusion Criteria:

* Current suicide or homicide risk
* Life-threatening or unstable medical condition
* Known or suspected prostate or chest cancer or history of polycythemia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Cutter, Ph.D., Study Director — Yale University; Declan T Barry, Ph.D., Principal Investigator — Yale University
Locations (1):
- MRU, APT Foundation, Inc, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Replacement: Testosterone replacement for hypogonadism.
  Testosterone replacement
- Waitlist Control: This arm involves watchful waiting.
  Waitlist control
Period: Overall Study
Arm/Group | Testosterone Replacement | Waitlist Control
Started | 8 | 7
Completed | 7 | 6
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Replacement | Waitlist Control | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10) | 48 (11) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Abstinence
Description: Number of participants who provided four consecutive weekly urines that were negative for illicit opioids in weeks 5 through 8.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Testosterone Replacement | Waitlist Control
Number analyzed (Participants) | 8 | 7
Participants | 5 | 4

2. Primary Outcome: Change in Pain Ratings
Description: Pain ratings will be assessed by self-report (4 items from Brief Pain Inventory). Change in pain ratings was assessed by examining the differences between pain ratings at baseline and week 8. Higher values are considered to be a worse outcome. The scale range is 0-10.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Testosterone Replacement | Waitlist Control
Number analyzed (Participants) | 8 | 7
units on a scale | 1.8 [.9 to 2.5] | 1.8 [1 to 2.6]

3. Primary Outcome: Change in Sexual Dysfunction From Baseline to Week 8
Description: Decreased sexual dysfunction will be assessed using the Erectile Function (EF) subscale of the International Index of Erectile Function (IIEF). The EF subscale has 6 items scored on a zero to five Likert-type scale. Change in sexual dysfunction was calculated by subtracting the mean EF subscale score at week 8 from the mean EF subscale score at baseline. The range of the EF subscale is 0-30 (with higher scores representing greater functioning). The Cut-offs for the EF subscales are as follows: no erectile dysfunction (score 26-30), mild erectile dysfunction (22-25), mild to moderate erectile dysfunction(17-21), moderate erectile dysfunction (11-16), and severe erectile dysfunction (0-10).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Replacement | Waitlist Control
Number analyzed (Participants) | 8 | 7
units on a scale | 6.95 (1.4) | -1 (1.3)

ADVERSE EVENTS:
Arm/Group | Testosterone Replacement | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Replacement (N=8) | Waitlist Control (N=7)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — patient reported general fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes